CLINICAL TRIAL: NCT00162799
Title: Phase IIa Study of Triflusal in the Attenuation of Insulin Resistance in Men and Woman With Obesity
Brief Title: Efficacy Pilot Study of Triflusal in the Attenuation of Insulin Resistance in Human Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: J. Uriach and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ICO5TRI/2/01
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2005-09

CONDITIONS: Insulin Resistance
Keywords: insulin resistance and inflamation; insulin sensitibity; obesity-induced insuline resistence; obesity-diabetes link; salicylate; insulin resistance in obesity health adults
MeSH Terms: conditions — Insulin Resistance | interventions — triflusal

INTERVENTIONS:
Drug: Triflusal (DCI)

SUMMARY:
To explore the efficacy of triflusal in the attenuation of insulin resistance in human obesity. Triflusal is a salicylate compound approved in several countries as antithrombotic agent (antiplatelet). The hypothesis is to explore if there is a reduction of obesity-induced insulin resistance by triflusal.

DETAILED DESCRIPTION:
Double-blind, randomized, cross-over (three periods) with two dose levels of triflusal, placebo-controlled.

Interventions: treatment periods Triflusal 600 mg/d, 15 days Triflusal 900 mg/d , 15 days placebo, 15 days

Washout period: 30 days

ELIGIBILITY:
Inclusion Criteria:

* Ages 35 to 60 years old

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2002-07; Study Completion 2004-12

PRIMARY OUTCOMES:
Increase of insulin sensitivity in apparently healthy men and woman evaluate by means of i.v. glucose tolerance test (PTEVGMR).

SECONDARY OUTCOMES:
Reduction antropometric measures associated with insulin resistance and arterial hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Manuel Fernández del Real, Dr, Principal Investigator — Unidad Diabetología. Serv Endocrino Hosp Josep Trueta
Locations (1):
- Unitat de Diabetologia, Endocrinologia y Nutrición Hosp Josep Trueta, Girona, Girona, Spain